CLINICAL TRIAL: NCT00081367
Title: Community-Based Cognitive Therapy for Suicide Attempters
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Gregory Brown, Research Associate Professor of Clinical Psychology in Psychiatry, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH067805 (NIH); R01MH067805 (NIH); DSIR 83-ATP
Record Dates: First submitted 2004-04-09; First posted 2004-04-12 (Estimated); Last update posted 2014-06-10 (Estimated); Status verified 2014-06

CONDITIONS: Suicide, Attempted
Keywords: Minority Groups
MeSH Terms: conditions — Suicide, Attempted

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive behavioral therapy (CBT) + standard care (Experimental): Participants will receive ten weekly sessions of treatment plus standard care for suicide prevention.
  Interventions: Behavioral: CBT; Behavioral: Standard care alone
- Standard care alone (Active Comparator): Participants will receive standard care for suicide prevention.
  Interventions: Behavioral: Standard care alone

INTERVENTIONS:
Behavioral: CBT — Participants will receive ten weekly sessions of treatment. Suicidal thoughts or attempts, hopelessness, depression, health care utilization, and overall psychological and social adaptation will be assessed.
  Arms: Cognitive behavioral therapy (CBT) + standard care
Behavioral: Standard care alone — Participants will receive standard care for suicide prevention.

SUMMARY:
This study will determine the effectiveness of cognitive behavioral therapy (CBT) in preventing future suicide attempts in repeat suicide attempters.

DETAILED DESCRIPTION:
Rates of mental health and substance use disorders are high among economically disadvantaged, ethnic minority populations. Studies have shown that CBT designed for this high-risk population is successful at reducing suicide attempts in people with suicidal thoughts or attempts. This study will implement a CBT intervention into the community and will focus on increasing compliance with psychiatric, substance abuse, and medical treatment.

Participants in this study will be randomly assigned to receive either CBT plus standard care or standard care alone. Participants who receive CBT will have ten weekly sessions of treatment. Suicidal thoughts or attempts, hopelessness, depression, health care utilization, and overall psychological and social adaptation will be assessed. Assessments will be made 1, 3, 6, 12, 18, and 24 months after study completion.

ELIGIBILITY:
Inclusion Criteria:

* Suicide attempt within 48 hours prior to being evaluated at the hospital
* English speaking
* Able to provide 2 verifiable contacts

Exclusion Criteria:

* Acute, unstable, or severe Axis III disorder or a severe Axis I disorder that may prevent safe participation in outpatient psychotherapy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2004-02; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Repeat suicide attempts | Measured during treatment and 1, 3, 6, 12, 18, and 24 months after study completion

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Brown GK, Ten Have T, Henriques GR, Xie SX, Hollander JE, Beck AT. Cognitive therapy for the prevention of suicide attempts: a randomized controlled trial. JAMA. 2005 Aug 3;294(5):563-70. doi: 10.1001/jama.294.5.563. PMID 16077050
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617